CLINICAL TRIAL: NCT07176143
Title: Study on the Clinical Efficacy and Safety of Infusing Human Bone Marrow Mesenchymal Stem Cells Via Uterine Artery for the Treatment of Infertility Due to Severe Intrauterine Adhesions
Brief Title: hBMSC Uterine Artery Infusion for Severe IUA-Related Infertility
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sixth Affiliated Hospital, Sun Yat-sen University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024ZSLYFEC-013
Record Dates: First submitted 2025-06-30; First posted 2025-09-16 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Intrauterine Adhesions
Keywords: intrauterine adhesions; uterine artery perfusion; human bone marrow mesenchymal stem cells
MeSH Terms: conditions — Gynatresia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stem cell therapy group (Experimental): Traditional hormone replacement cycle therapy was used (estrogen Valerate tablets 3mg bid for 28 days, followed by Dydrogesterone tablets 10mg bid for the last 10 days of the 28 day period) + hBMSC infusion via uterine artery.
  Interventions: Procedure: Delivering human bone marrow mesenchymal stem cells via the uterine artery
- Control group (No Intervention): Traditional hormone replacement cycle therapy was used (estrogen Valerate tablets 3mg bid for 28 days, followed by Dydrogesterone tablets 10mg bid for the last 10 days of the 28 day period).

INTERVENTIONS:
Procedure: Delivering human bone marrow mesenchymal stem cells via the uterine artery — Interventional Uterine Artery Infusion of Human Bone Marrow Mesenchymal Stem Cells (hBMSCs):
  Subjects in the experimental group will undergo iodine allergy testing and groin area shaving/disinfection preoperatively. The procedure is performed on Day 10 of the endometrial proliferation phase.
  Step-by-Step Procedure:
  1. Positioning & Anesthesia: (Patient placed in supine position; Local infiltration anesthesia administered)
  2. Arterial Access: (Femoral artery punctured using Seldinger technique; Vascular sheath and catheter inserted)
  3. Catheterization: (Catheter/microcatheter advanced into one uterine artery; Position confirmed by angiography)
  4. Stem Cell Infusion: (Under fluoroscopic guidance, slowly inject 15mL solution containing 1×10⁶ cells/kg hBMSCs via microcatheter)
  5. Postoperative Care: (Hospital observation for 48 hours)
  6. Concurrent Treatment: (Hormone replacement therapy cycle maintained during the procedure month)
  Treatment Frequency: Single intervention
  Other Names: Arterial perfusion of bone marrow mesenchymal stem cells
  Arms: Stem cell therapy group

SUMMARY:
The goal of this clinical trial is to test a new approach: delivering human bone marrow mesenchymal stem cells (hBMSCs) via the uterine artery to treat infertility caused by severe intrauterine adhesions (IUA). This method may help stem cells better reach the deep layer of the endometrium, promote endometrial repair, and improve pregnancy chances.

Primary Objective: To assess whether stem cell therapy improves pregnancy success rates (clinical pregnancy rate after embryo transfer) in infertility patients with severe IUA undergoing IVF.

Secondary Objectives:

1. To evaluate the safety of stem cell therapy (e.g., side effects or complications).
2. To explore how stem cells help repair the endometrium (e.g., by promoting endometrial growth or improving uterine conditions).

By tracking endometrial thickness, embryo implantation rate, clinical pregnancy rate, and other indicators, we will evaluate whether this new approach is safe and effective.

Treatment Groups:

Control group: Standard hormone replacement therapy (HRT) cycle medication only.

Stem cell therapy group: Standard HRT medication + hBMSC infusion via uterine artery.

Both groups will undergo embryo transfer, and clinical pregnancy rates will be compared.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects fully comprehend the screening process and study objectives, demonstrate adequate understanding of and compliance with the trial protocol, and provide signed informed consent.
2. Age between 20 and 38 years.
3. Body mass index (BMI) 18-27 kg/m².
4. Regular menstrual cycles (27-35 days) for ≥6 months.
5. Normal ovarian reserve: Antral follicle count (AFC) ≥6; Follicle-stimulating hormone (FSH) 1-10 IU/L on cycle days 2-4; Baseline sex hormones within normal laboratory ranges.
6. Negative serology within 6 months for: HIV antibodies; Treponema pallidum antibodies (TPA); Hepatitis B surface antigen (HBsAg); Hepatitis C virus antibodies (HCV-Ab).
7. ≥2 good-quality blastocysts (D5/D6) according to Gardner grading criteria.
8. Prior hysteroscopic diagnosis of severe intrauterine adhesions (IUA) treated with electroresection, with normal uterine cavity morphology confirmed by hysteroscopy within 3 months.
9. History of canceled frozen embryo transfers due to persistently thin endometrium (<6 mm) in HRT and/or natural cycles during the late proliferation phase.

Exclusion Criteria:

1. Ovarian cysts ≥20 mm, submucosal/intramural uterine fibroids >30 mm, pituitary tumors, or malignancy in any organ.
2. Clinically significant uterine (endometrial polyps, IUA, malformations, endometriosis) or adnexal (hydrosalpinx) abnormalities.
3. Recurrent implantation failure (≥3 consecutive transfers with ≥6 good-quality embryos failing).
4. Unexplained abnormal vaginal bleeding.
5. Active pelvic inflammatory disease.
6. Reproductive tract malformations incompatible with pregnancy.
7. Abnormal cervical cytology (TCT) within 1 year before screening.
8. Severe hepatic/renal impairment, cardiac disease, or hypertension.
9. History of thrombophlebitis or thromboembolism.
10. Platelet count <100×10⁹/L, hemoglobin <100 g/L, or hematologic disorders (e.g., idiopathic thrombocytopenic purpura).
11. Clinically significant systemic diseases (e.g., diabetes, tuberculosis).
12. History of recurrent miscarriage.
13. Chromosomal abnormalities in either partner.
14. Genetic disorders (per Maternal and Infant Health Care Law) contraindicating pregnancy in either partner.
15. Exposure to teratogenic radiation, toxins, or medications in either partner.
16. Participation in other drug/device trials within 3 months prior to enrollment.
17. Any condition (comorbidity, surgery, medication, or abnormal lab results) deemed by investigators to affect trial outcomes.
18. Inability or refusal to comply with protocol requirements (including scheduled visits and tests).

Ages: 20 Years to 38 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-09-30 (Estimated); Primary Completion 2027-12-30 (Estimated); Study Completion 2028-12-30 (Estimated)

PRIMARY OUTCOMES:
Clinical pregnancy rate | 90 days
  To assess whether stem cell therapy improves pregnancy success rates (clinical pregnancy rate after embryo transfer) in infertility patients with severe IUA undergoing IVF.

SECONDARY OUTCOMES:
Safety of transuterine arterial infusion of hBMSCs | 6 month
  Immediate adverse events include monitoring for infusion-related reactions such as fever, chills, allergic manifestations, local pain at the uterine artery puncture site or pelvis, and hemodynamic instability. Within the first week, short-term safety evaluation emphasizes detecting infection markers, thrombotic complications, and bleeding risks. Medium-term safety (1-3 months) involves assessing hepatic/renal function abnormalities, potential immune responses through autoantibody testing and lymphocyte profiling, and imaging surveillance for ectopic tissue formation. Long-term follow-up (≥6 months) systematically evaluates tumorigenic risks through serum tumor markers and pelvic imaging, screens for endometrial malignant transformation via biopsy, and monitors ovarian reserve through hormonal (FSH, AMH) and follicular tracking.
Exploration of related mechanisms | 1 year
  Exploring the mechanism of endometrial proliferation in infertile subjects with severe intrauterine adhesions treated by infusion of human bone marrow mesenchymal stem cells via uterine artery.

IPD SHARING:
Plan to Share IPD: No